CLINICAL TRIAL: NCT01236105
Title: Evaluation of the Impact of Activated Charcoal and Time of Dose on the Absorption of LY2624803 in Healthy Subjects
Brief Title: Effect of Activated Charcoal and Time of Dose on the Pharmacokinetics of LY2624803 in Healthy Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 12814; I2K-MC-ZZBQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Results first posted 2011-12-22 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-11

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Charcoal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 6 mg LY2624803 Alone Morning Dosing (Experimental): Participants received 6 milligrams (mg) LY2624803 alone orally (po) at approximately 0800 hours following an overnight fast.
  Interventions: Drug: LY2624803
- 6 mg LY2624803 Morning Dosing + Activated Charcoal (Experimental): Participants received 6 mg LY2624803 po at approximately 0800 hours following an overnight fast, followed 1 hour later by a single po dose of 1 gram per kilogram (g/kg) body weight of activated charcoal, mixed with caffeine-free diet cola.
  Interventions: Drug: LY2624803; Other: Activated Charcoal
- 6 mg LY2624803 Alone Evening Dosing (Experimental): Participants received 6 mg LY2624803 alone po at approximately 2200 hours following a 4-hour fast.
  Interventions: Drug: LY2624803

INTERVENTIONS:
Drug: LY2624803 — Administered orally (po), once.
Other: Activated Charcoal — Administered po
  Arms: 6 mg LY2624803 Morning Dosing + Activated Charcoal

SUMMARY:
The purpose of this study is to determine the effect of activated charcoal and dosing time on the absorption of LY2624803 in healthy subjects. In this crossover study, there are three treatments with a washout period of at least 7 days in between treatments. Each subject will participate in all three treatments with random assignment to the treatment sequence.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination.
* Male subjects with female partners of child-bearing potential and female subjects of child-bearing potential, agree to use 2 reliable methods of contraception from the time of the first dose until 3 months after the last dose of study drug or are women not of child-bearing potential due to postmenopausal or permanently sterilized [for example, tubal occlusion, hysterectomy, bilateral salpingectomy]).
* Have a body mass index (BMI) between 18.5 and 32 kilograms per square meter (kg/m2), inclusive, and a body weight of 50 kg or above at screening.
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have venous access sufficient to allow blood sampling as per the protocol.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Have given written informed consent approved by Lilly and the ethical review board governing the site.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 90 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device (other than the study drug used in this study), or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies to LY2624803 or related compounds.
* Are persons who have previously completed or withdrawn from this study or any other study investigating LY2624803.
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Have an abnormal blood pressure as determined by the investigator.
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal (except appendectomy), endocrine, hematological, dermatological, venereal, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, of constituting a risk when taking the study medication, or of interfering with the interpretation of data.
* Show evidence or history of postural hypotension, loss of consciousness, explained or unexplained syncope or seizure episodes or a family history of seizures. A history of a single febrile convulsion is acceptable.
* Show evidence of significant active neuropsychiatric disease.
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Are women with a positive pregnancy test or women who are lactating.
* Intend to use over-the-counter or prescription medications, with the exception of vitamins and paracetamol, which cannot be safely discontinued within 7 days prior to admission.
* Have donated blood of more than 500 milliliters (mL) within the last 3 months prior to screening.
* Have an average weekly alcohol intake that exceeds 28 units per week (males) and 21 units per week (females), and are subjects unwilling to stop alcohol consumption from 48 hours prior to admission until discharge from the unit for each treatment period, and to limit alcohol intake to a maximum of 2 units/day between treatment periods.
* Have a history of breast cancer.
* Are subjects with excessive xanthine consumption.
* Exhibit any other condition, which, in the opinion of the investigator would preclude participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2624803: Participants received each of the following 3 study treatments:
  LY2624803 Alone Morning Dosing: Participants received 6 milligrams (mg) LY2624803 alone, orally (po) once at approximately 0800 hours following an overnight fast.
  LY2624803 Morning Dosing Plus Activated Charcoal: Participants received 6 mg LY2624803 po once at approximately 0800 hours following an overnight fast, followed 1 hour later by a single po dose of 1 gram per kilogram (g/kg) body weight of activated charcoal, mixed with caffeine-free diet cola.
  LY2624803 Alone Evening Dosing: Participants received 6 mg LY2624803 alone po once at approximately 2200 hours following a 4-hour fast.
Period: Overall Study
Arm/Group | LY2624803
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LY2624803
Number analyzed (Participants) | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 32.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20
  Black | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 21

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve (AUC) for LY2624803 and the Metabolite LSN2797276
Description: AUC from time 0, extrapolated to infinity, estimated for both LY2624803 and the metabolite LSN2797276.
Time Frame: Predose and up to Day 4
Population: All participants who received at least 1 dose of LY2624803 and have evaluable pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Groups:
- LY2624803 Alone Morning Dosing: Participants received 6 milligrams (mg) LY2624803 alone, orally (po) once (QD) at approximately 0800 hours following an overnight fast.
- LY2624803 Morning Dosing Plus Activated Charcoal: Participants received 6 mg LY2624803 po QD at approximately 0800 hours following an overnight fast, followed 1 hour later by a single po dose of 1 gram per kilogram (g/kg) body weight of activated charcoal, mixed with caffeine-free diet cola.
- LY2624803 Alone Evening Dosing: Participants received 6 mg LY2624803 alone po QD at approximately 2200 hours following a 4-hour fast.
Arm/Group | LY2624803 Alone Morning Dosing | LY2624803 Morning Dosing Plus Activated Charcoal | LY2624803 Alone Evening Dosing
Number analyzed (Participants) | 21 | 20 | 21
nanogram*hour per milliliter (ng*h/mL)
  LY2624803 | 5240 (30) | 3340 (30) | 4620 (30)
  LSN2797276 (N=18, 12, 15) | 192 (23) | 112 (19) | 188 (26)

2. Primary Outcome: Maximum Concentration (Cmax) for LY2624803 and the Metabolite, LSN2797276,
Description: Cmax estimated for both LY2624803 and the metabolite LSN2797276.
Time Frame: Predose and up to Day 4
Population: All participants who received at least 1 dose of LY2624803 and have evaluable pharmacokinetic (PK) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | LY2624803 Alone Morning Dosing | LY2624803 Morning Dosing Plus Activated Charcoal | LY2624803 Alone Evening Dosing
Number analyzed (Participants) | 21 | 20 | 21
nanogram per milliliter (ng/mL)
  LY2624803 | 368 (26) | 335 (35) | 273 (17)
  LSN2797276 | 6.22 (27) | 5.11 (41) | 5.94 (28)

3. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) for LY2624803 and the Metabolite, LSN2797276
Description: Tmax, estimated for both LY2624803 and the metabolite LSN2797276.
Time Frame: Predose and up to day 4
Population: All participants who received at least 1 dose of LY2624803 and have evaluable pharmacokinetic (PK) data.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | LY2624803 Alone Morning Dosing | LY2624803 Morning Dosing Plus Activated Charcoal | LY2624803 Alone Evening Dosing
Number analyzed (Participants) | 21 | 20 | 21
hours (h)
  LY2624803 | 1.50 [0.50 to 2.50] | 0.75 [0.50 to 1.50] | 2.00 [1.50 to 6.00]
  LSN2797276 | 4.00 [2.00 to 8.00] | 4.00 [0.75 to 6.03] | 8.00 [2.00 to 12.00]

ADVERSE EVENTS:
Groups:
- LY2624803 Morning Dosing: LY2624803 Alone Morning Dosing: Participants received 6 milligrams (mg) LY2624803 alone, orally (po) once at approximately 0800 hours following an overnight fast.
- LY2624803 Morning Dosing + Activated Charcoal: LY2624803 Morning Dosing Plus Activated Charcoal: Participants received 6 mg LY2624803 po once at approximately 0800 hours following an overnight fast, followed 1 hour later by a single po dose of 1 gram per kilogram (g/kg) body weight of activated charcoal, mixed with caffeine-free diet cola.
- LY2624803 Evening Dosing: LY2624803 Alone Evening Dosing: Participants received 6 mg LY2624803 alone po once at approximately 2200 hours following a 4-hour fast.
Arm/Group | LY2624803 Morning Dosing | LY2624803 Morning Dosing + Activated Charcoal | LY2624803 Evening Dosing
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 13/21 | 8/21 | 10/21
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2624803 Morning Dosing (N=21) | LY2624803 Morning Dosing + Activated Charcoal (N=21) | LY2624803 Evening Dosing (N=21)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days